CLINICAL TRIAL: NCT03191708
Title: Functional Diagnostic Accuracy of Quantitative Flow Ratio in On-line Assessment of Coronary Stenosis (The FAVOR II China Study)
Brief Title: The FAVOR II China Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Pulse Medical Imaging Technology (Shanghai) Co., Ltd (Industry)
Responsible Party: Principal Investigator, fuwaihospital, Professor, China National Center for Cardiovascular Diseases
Other Study IDs: FAVOR II -1608
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Disease; Arterial Occlusive Diseases; Heart Diseases; Vascular Diseases
Keywords: Fractional Flow Reserve; Quantitative Coronary Angiography; Coronary artery disease; Angina pectoris; Quantitative Flow Ratio
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Disease; Arterial Occlusive Diseases; Heart Diseases; Vascular Diseases; Angina Pectoris | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve (FFR) — FFR measured by pressure wire, QFR computed by coronary angiographic images
  Other Names: Quantitative Flow Ratio (QFR)

SUMMARY:
Quantitative Flow Ratio (QFR) is a novel method for evaluating the functional significance of coronary stenosis. The purpose of the FAVOR II China study is to evaluate the diagnostic accuracy of on-line QFR with FFR as the reference standard. The secondary purpose is to compare the diagnostic accuracies between online QFR and online QCA, with FFR as the reference standard.

DETAILED DESCRIPTION:
Patients at high risk of having one or more coronary stenosis are evaluated routinely by invasive coronary angiography. Lesions are often quantified by QCA, but fractional flow reserve is increasingly used to assess functional significance of identified stenosis. FFR is assessed during CAG by advancing a wire with a pressure transducer towards the stenosis and measure the ratio in pressure between the two sides of the stenosis during medical induced maximum blood flow (hyperemia).

The solid evidence for FFR evaluation of coronary stenosis and the relative simplicity in performing the measurements have supported adoption of an FFR based strategy in many centers but the need for interrogating the stenosis by a pressure wire, the cost of the wire, and the drug inducing hyperemia limits more widespread adoption.

QFR is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on two angiographic projections. The FAVOR Pilot study (Tu et al.) showed promising results for core laboratory QFR analysis in selected patients. However, the accuracy of QFR when assessed online in the catheterization laboratory is unknown. The purpose of the FAVOR II China study is to evaluate the diagnostic accuracy of on-line QFR with FFR as the reference standard. The secondary purpose is to compare the diagnostic accuracies between online QFR and online QCA, with FFR as the reference standard. It is a prospective and multi-center trial with a total of 308 patients conducted at 5 Chinese centers.

ELIGIBILITY:
Inclusion Criteria:

General Criteria:

* Stable and unstable angina pectoris or secondary evaluation of stenosis after acute MI
* Age > 18 years
* Able to provide signed informed consent

Angiographic inclusion criteria:

* At least one stenosis with diameter stenosis of 30%-90% by visual estimate
* Reference vessel size > 2 mm in stenotic segment by visual estimate

Exclusion Criteria:

General Criteria:

* Ineligible for diagnostic intervention or FFR examination
* Myocardial infarction within 72 hours
* Severe heart failure (NYHA≥III)
* S-creatinine>150µmol/L or GFR<45 ml/kg/1.73m2
* Allergy to contrast agent or adenosine
* Factors that might substantially impact the angiographic image quality, e.g, frequent atrial premature beat or atrial fibrillation

Angiographic exclusion criteria:

* The interrogated stenosis is caused by myocardial bridge
* Ostial lesions less than 3 mm to the aorta
* Side branches of the bifurcation lesions with Median Classification of 111 or 101
* Poor angiographic image quality precluding contour detection
* Severe overlap of stenotic segments
* Severe tortuosity of target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease admitted for coronary angiography due to high risk of significant coronary stenosis
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of online QFR to determine presence or absence of hemodynamically-significant coronary artery stenosis at the vessel level using binary outcomes when compared to FFR as the reference standard. | 1 hour
  Presence of hemodynamically-significant coronary artery stenosis : FFR <= 0.80.

SECONDARY OUTCOMES:
In comparison to online 2D QCA, sensitivity and specificity of online QFR to determine presence or absence of hemodynamically-significant coronary artery stenosis at the vessel level using binary outcomes when compared to FFR as the reference standard | 1 hour
  Sensitivity: Proportion of patients with positive QFR of FFR positive patients (true positives) compared to proportion of patients with positive percentual diameter stenosis (DS%) assessed by 2D QCA of FFR positive patients (true positives).
  Specificity: Proportion of patients with negative QFR of FFR negative patients (true negatives) compared to proportion of patients with negative DS% assessed by 2D QCA of FFR negative patients (true negatives).
The numerical difference between online QFR and core lab QFR. | 1 hour
The numerical difference between online QFR and FFR. | 1 hour
The area under the receiver operating characteristic curve of online QFR in determining presence or absence of hemodynamically-significant coronary artery stenosis at the vessel level using binary outcomes when compared to FFR as the reference standard | 1 hour
  Presence of hemodynamically-significant coronary artery stenosis : FFR <= 0.80.
Feasibility of online computation of QFR | 1 hour
  Percentage of successful QFR in all vessels sent to QFR computation

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Guangdong General Hospital, Guangzhou
  - Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai

REFERENCES:
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Derived] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020